CLINICAL TRIAL: NCT02439177
Title: Evaluating System Accuracy and User Performance of Omnitest® Blood Glucose Monitoring Systems for Self-testing in Managing Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPM-G-V-1503
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes
Keywords: Blood glucose monitoring system; System Accuracy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omnitest 3 (Experimental): Blood glucose monitoring system
  Interventions: Device: Blood glucose monitoring system (Omnitest 3)
- Omnitest 5 (Experimental): Blood glucose monitoring system
  Interventions: Device: Blood glucose monitoring system (Omnitest 5)

INTERVENTIONS:
Device: Blood glucose monitoring system (Omnitest 3)
  Arms: Omnitest 3
Device: Blood glucose monitoring system (Omnitest 5)
  Arms: Omnitest 5

SUMMARY:
The aim of this study is to determine the System Accuracy and User Performance evaluation of the mentioned BGM systems by gaining a sufficient amount of measured data from capillary blood.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with type 1 or type 2 diabetes, for the evaluation of System Accuracy also healthy subjects
* Age ≥ 18
* Signed and dated informed consent form
* For small modifications of the insulin doses to achieve certain blood glucose values (System Accuracy evaluation): Male or female subjects with diabetes mellitus type 1 with intensified insulin therapy (intensified conventional therapy - I.C.T.) or insulin pump therapy (continuous subcutaneous insulin infusion - C.S.I.I.)

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute illness that, in the opinion of the investigating physician, might confound the results of the test or which could result in a risk to the subject caused by the test.
* Severe chronic illness besides Diabetes mellitus as assessed by the investigating physician that might confound the results of the test or which could result in a risk to the subject caused by the test.
* Mental incapacity or language barriers precluding adequate compliance with the test procedures
* Legal incompetence or limited legal competence
* Dependency from the Sponsor or the clinical Investigator (e.g. co-workers of the Sponsor or the clinical research centre)
* For User Performance evaluation: Subjects having participated in a study with Omnitest® 5 before.
* For System Accuracy evaluation: subjects intended to provide blood samples with glucose concentrations between 50 and 80 mg/dl must not have coronary heart disease, myocardial infarction in history, cerebral events in history, peripheral artery occlusive disease or impaired hypoglycaemia awareness
* Anamnestically relevant amounts of interfering substances in the blood, following labelling in the instructions for use as reviewed and evaluated by a physician during screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
System accuracy, results obtained from fingertip using blood glucose monitoring systems compared to a reference equipment | up to 7 hours
User Performance of blood glucose monitoring system indicated by patient | up to 7 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany